CLINICAL TRIAL: NCT02784587
Title: Feasibility of Perioperative Stellate Ganglion Blocks in Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Christopher Connors, MD (Other)
Responsible Party: Sponsor-Investigator, Christopher Connors, MD, Staff Anesthesiologist, MaineHealth
Organization: MaineHealth (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: #4624
Record Dates: First submitted 2016-05-17; First posted 2016-05-27 (Estimated); Results first posted 2019-07-08 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-04

CONDITIONS: Atrial Fibrillation
Keywords: stellate ganglion block; cardiac surgery
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Stellate Ganglion Block (Experimental): All patients in the study will receive a stellate ganglion block in order to asses the feasibility and efficacy of this procedure performed by cardiac anesthesiologists in the operating room.
  Interventions: Procedure: Stellate Ganglion Block

INTERVENTIONS:
Procedure: Stellate Ganglion Block — After induction of general anesthesia, patients will receive a stellate ganglion block using a standard and well described paratracheal technique, which typically requires about 3 minutes to perform. The patient's head will be extended and a 4-5-cm, 22-gauge needle inserted at the medial edge of the sternocleidomastoid muscle just below the level of the cricoid cartilage at the level of the transverse process of C6 (Chassaignac's tubercle) or C7 (3-5 cm above the clavicle). The non-operative hand will retract the muscle together with the carotid sheath prior to needle insertion. After advancing to the transverse process the needle will be withdrawn 2-3 mm prior to injection. A negative aspiration test will be performed in two planes before a 1-ml test dose is used to exclude unintentional intravascular injection (vertebral or subclavian arteries) or subarachnoid injection into the dural sleeve.4 A total of 10 ml of 0.25% bupivacaine will be injected.

SUMMARY:
Based upon Northern New England Cardiovascular Study Group data, the rate of post operative atrial fibrillation (POAF) requiring treatment following coronary artery bypass grafting (CABG) at Maine Medical Center (MMC) is currently 30%. Nationally, POAF occurs in up to 40% of patients post CABG, 50% of patients after valve surgery, 64% of patients post mitral valve and CABG and 49% after aortic valve replacement. Atrial fibrillation worsens a patient's hemodynamic status and increases the risk of congestive heart failure (CHF), embolic events and longer ICU stays leading to increased patient morbidity and strain on financial resources. In the U.S., POAF carries a higher risk of stroke (37% OR 2.0 in-hospital mortality (OR = 1.7), worsened survival (74% versus 87%), and an additional 4.9 days and $10,000-$11,500 in hospital stay costs.

Atrial fibrillation requires both an initiation trigger and favorable environment for maintenance and the sympathetic and parasympathetic nervous systems play important roles in this regard. Unfortunately, the precise mechanisms of POAF are still being investigated. This postoperative complication has persisted in spite of efforts to mitigate it pharmacologically with beta blockers and amiodarone, an experience shared by most other cardiac surgery centers.

The stellate ganglion is formed by the fusion of the inferior cervical sympathetic ganglion and first thoracic sympathetic ganglion. By modulating the sympathetic component of the autonomic nervous system, stellate ganglion stimulation has been shown to facilitate induction of atrial fibrillation while ablation may reduce or prevent episodes. Human studies have further supported this model.

Preliminary studies of perioperative stellate ganglion block (SGB) in cardiac surgery suggest that this technique may reduce or prevent episodes of POAF requiring treatment. The investigator's ultimate goal is to determine whether SGB reduces the incidence of POAF in specific cardiac surgery populations at MMC. First, however, the investigator proposes to test the hypothesis that SGB, performed perioperatively by cardiac anesthesiologists in a population of patients undergoing cardiac surgery, is both safe and clinically feasible.

DETAILED DESCRIPTION:
Patients at MMC undergoing transapical transcatheter aortic valve replacement (TA TAVR) routinely receive a paravertebral block for analgesia. This has the added benefit of providing a unilateral sympathectomy which may be analogous to a stellate ganglion block, albeit via a different technique. In a recent retrospective chart review, TA TAVR block patients showed a decreased rate of new onset POAF. Furthermore, when studying whether pre-emptive stellate ganglion block increases the patency of radial artery grafts in coronary bypass surgery, researchers found a statistically significant decrease (p = 0.048) in atrial fibrillation and the use of anti-arrhythmic agents. Unfortunately, this was a secondary outcome in a small patient population and, while suggestive, the study was not sufficiently powered to draw a definitive conclusion. Importantly, however, they reported no complications related to the block in the fifty patients who received an intervention. Lastly, an additional study demonstrated the safety and feasibility of stellate ganglion mapping and ablation during CABG while also suggesting a clinically significant effect on POAF, but used a permanent, technically complex and time intensive procedure.

The investigator's hypothesis is that perioperative SGB in cardiac surgery is clinically efficient and efficacious. To address this, the investigator will:

1. Recruit 49 patients to undergo perioperative SGB during prior to cardiac surgery (CABG, CABG/Aortic Valve Replacement, Aortic Valve Replacement).
2. Monitor the safety of SGB using post procedure surface ultrasound of the neck and active solicitation on Post-op Day (POD) 0 and 1 for identified complications, in addition to routine clinical monitoring.
3. Assess clinical feasibility of SGB by measuring procedural efficacy and efficiency:

   1. Efficacy will be measured using post procedure hand temperature; success is indicated by an increase greater than 1 degree Celsius.
   2. Efficiency will be measured as the time to complete the block and the time added to the standard anesthesia induction sequence, as a proportion of total time in the operating room.

Significance: If the investigator is able to demonstrate that perioperative SGB in cardiac surgery is safe and clinically feasible, the next step will be to design a study to investigate the effect of SGB on POAF incidence (and thereby its attendant morbidity, mortality and costs) in this clinical population.

ELIGIBILITY:
Inclusion Criteria:

* scheduled for AVR, CABG, or CABG/AVR

Exclusion Criteria:

* age <18 years
* pregnant women
* prisoners
* patients having emergency surgery
* patients with any clinical contraindication to SGB, including: amide local anesthetic allergy or hypersensitivity, carotid vascular disease as defined by ipsilateral prior carotid endarterectomy or carotid stent, superficial infection at the proposed puncture site, contralateral phrenic or laryngeal nerve palsies
* patients with severe chronic obstructive pulmonary disease as defined by the need for home oxygen
* patients who do not speak or write English or are unable to give informed consent
* patients with a history of atrial fibrillation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-05-31 (Actual); Primary Completion 2016-12-06 (Actual); Study Completion 2016-12-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Connors, MD, Principal Investigator — MaineHealth

RESULTS

PARTICIPANT FLOW:
Groups:
- Stellate Ganglion Block: All patients in the study will receive a stellate ganglion block in order to asses the feasibility and efficacy of this procedure performed by cardiac anesthesiologists in the operating room.
  Stellate Ganglion Block: After induction of general anesthesia, patients will receive a stellate ganglion block using a standard and well described paratracheal technique, which typically requires about 3 minutes to perform. The patient's head will be extended and a 4-5-cm, 22-gauge needle inserted at the medial edge of the sternocleidomastoid muscle just below the level of the cricoid cartilage at the level of the transverse process of C6 (Chassaignac's tubercle) or C7 (3-5 cm above the clavicle). The non-operative hand will retract the muscle together with the carotid sheath prior to needle insertion. After advancing to the transverse process the needle will be withdrawn 2-3 mm prior to injection.
Period: Overall Study
Arm/Group | Stellate Ganglion Block
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Stellate Ganglion Block: All patients in the study will receive a stellate ganglion block in order to asses the feasibility and efficacy of this procedure performed by cardiac anesthesiologists in the operating room.
  Stellate Ganglion Block: After induction of general anesthesia, patients will receive a stellate ganglion block using a standard and well described paratracheal technique, which typically requires about 3 minutes to perform. The patient's head will be extended and a 4-5-cm, 22-gauge needle inserted at the medial edge of the sternocleidomastoid muscle just below the level of the cricoid cartilage at the level of the transverse process of C6 (Chassaignac's tubercle) or C7 (3-5 cm above the clavicle). The non-operative hand will retract the muscle together with the carotid sheath prior to needle insertion.
Arm/Group | Stellate Ganglion Block
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 22
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Success of Stellate Ganglion Block
Description: Correct placement of stellate ganglion block as measured by a temperature rise of at least 1 degree Celsius in the ipsilateral hand
Time Frame: day of surgery
Measure: Count of Participants; unit: Participants
Groups:
- Stellate Ganglion Block: All patients in the study will receive a stellate ganglion block in order to asses the feasibility and efficacy of this procedure performed by cardiac anesthesiologists in the operating room.
  Stellate Ganglion Block: After induction of general anesthesia, patients will receive a stellate ganglion block using a standard and well described paratracheal technique, which typically requires about 3 minutes to perform. The patient's head will be extended and a 4-5-cm, 22-gauge needle inserted at the medial edge of the sternocleidomastoid muscle just below the level of the cricoid cartilage at the level of the transverse process of C6 (Chassaignac's tubercle) or C7 (3-5 cm above the clavicle).
Arm/Group | Stellate Ganglion Block
Number analyzed (Participants) | 25
Participants | 22

2. Secondary Outcome: Rate of Atrial Fibrillation
Description: The current rate of atrial fibrillation is measured by the Northern New England Cardiac Database, this existing database will track a-fib rates until the patients are discharged from the hospital after surgery.
Time Frame: Through study completion, approximately 1 year
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Patients were monitored for adverse events until discharged from the hospital, at least 3 days post-operatively.
Arm/Group | Stellate Ganglion Block
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No